CLINICAL TRIAL: NCT02382614
Title: Safety and Effectiveness of the Spiration Valve System (SVS) in Air Leaks
Brief Title: Spiration Valves Against Standard Therapy
Acronym: VAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: business reasons
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Air Leaks
Keywords: Endobronchial Valve; Minimally Invasive; Intrabronchial Valves; Digital Thoracic Drainage System; Spiration Valve System; Prolonged Air Leak; Persistent Air Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spiration Valve System (Experimental): The treatment group will have valves deployed to achieve leak isolation.
  Interventions: Device: Spiration Valve System
- Medical Management (No Intervention): The control group for this study will receive standard chest tube drainage management and standard-of-care interventions. This group will be evaluated and followed in the same manner as the treatment group, but without having valves placed.

INTERVENTIONS:
Device: Spiration Valve System
  Arms: Spiration Valve System

SUMMARY:
VAST is a multicenter, prospective, randomized, controlled study designed to evaluate treatment of persistent air leak with the SVS as compared to standard chest tube drainage management and other standard-of-care interventions in the control group. Eligible subjects will be randomized to receive either Spiration Valves (investigational arm) or continue standard-of-care treatment (control arm). Once the air leak has resolved, Spiration Valves should be removed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an air leak ≥ 100 mL/min, as measured by a digital thoracic drainage system (DTDS)
* Subject has air leak present on at least the 5th day following origination.

Exclusion Criteria:

* Subject has air leak only on forced exhalation or cough
* Subject has sepsis
* Subject has pneumonia
* Subject has Acute Respiratory Distress Syndrome (ARDS)
* Subject is not an appropriate candidate for, or unable to tolerate, flexible bronchoscopy procedures
* Subject has undergone a bone marrow transplant
* Subject has a primary pneumothorax
* Subject has undergone a prior intervention (including pleurodesis, surgery, blood patch, and pneumoperitoneum) or valve placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-05; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Time to Air Leak Cessation | Two weeks

OTHER OUTCOMES:
Incidence of SAE | Six weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - El Camino Hospital, Mountain View, California
  - California Pacific Medical Center, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Southern Illinois University, Springfield, Illinois
  - Olathe Medical Center, Olathe, Kansas
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dartmouth Mary Hitchcock Memorial Hospital, Hanover, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Medical Center, Seattle, Washington